CLINICAL TRIAL: NCT05065346
Title: A Study to Evaluate the Efficacy of Neoadjuvant DaRT for Locally Advanced Oral Cavity Squamous Cell Carcinoma
Brief Title: Neoadjuvant DaRT for Locally Advanced Oral Cavity SCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-OCC-00
Record Dates: First submitted 2021-09-12; First posted 2021-10-04 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma
Keywords: Oral Cavity Squamous Cell Carcinoma; Radiotherapy; Brachytherapy; Alpha Radiation
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device (DaRT) as a treatment prior to additional radiation or chemo therapy.

DETAILED DESCRIPTION:
The study is planned as a phase II, single arm interventional, open-label, multi-center, prospective study evaluating DaRT as a neoadjuvant therapy in patients with advanced oral cavity Squamous Cell Carcinoma.

The study will enroll 79 subjects with pathologically confirmed, previously untreated, resectable squamous cell carcinoma of the oral cavity above the age of 18.

This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

The target lesion will be inserted with DaRT in a neo-adjuvant setting. DaRT seeds will be removed 15 days following the insertion. Surgery will follow 15 to 20 days after removal of the DaRT seeds followed by standard chemoradiotherapy or radiotherapy alone based on histopathology.

The primary outcome of the study will be the assessment of the major pathological response.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed, previously untreated, resectable squamous cell carcinoma of the oral cavity (no involvement of the lips);
2. T1-T2, N1-N2; T3 N0-2 with T3 <5 cm, depth of infiltration <15 mm, (AJCC version 8 oral cavity);
3. Tumor must be potentially curable by conventional methods;
4. Primary tumor must be amenable for complete coverage (including margins) by the DaRT seeds;
5. Assessment by a Multi-Disciplinary Team (MDT) of the treatment naïve patient and suitable for DaRT based on diagnostic, contrast enhanced whole body PET-CT - and MRI at the discretion of the investigator - within 2 weeks prior to enrolment. MDT preferably composed of a head and neck/ear, nose, and throat (ENT) surgeon, medical oncologist, radiologist, radiotherapist, and pathologist but at least a surgeon and a radiotherapist;
6. Age 18 and older;
7. Eastern Cooperative Oncology Group (ECOG)/ World Health Organization (WHO) Performance status 0-2;
8. Adequate bone marrow function as demonstrated by neutrophils (ANC) ≥ 1,5 109 /L, platelet count ≥ 100 109 /L, leukocytes (WBC) ≥ 3.0 109 /L;
9. Hemoglobin ≥ 9.0 g/dL
10. Calculated creatinine clearance (CL) > 60 mL/min by the Cockcroft-Gault formula;
11. Coagulation parameter (as per institution's standard international normalized ratio (INR), PT or Quick PT) is within the normal ranges, or within the expected target range of their current dose for those patients receiving anticoagulant therapy.
12. Women of child-bearing potential (WOCBP) must have a negative serum pregnancy test within 21 days prior to the DaRT insertion.

    Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e. females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antioestrogens, low body weight, ovarian suppression or other reasons.
13. Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last dose of treatment.

    Note: A highly effective method of birth control is defined as a method which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:
    * Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
    * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
    * Intrauterine device (IUD)
    * Intrauterine hormone-releasing system (IUS)
    * Bilateral tubal occlusion
    * Vasectomized partner
    * Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
14. Female subjects who are breast-feeding should discontinue nursing prior to starting treatment and until 6 months after the last dose of study treatment;
15. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up;
16. Willing and able to provide tumor specimen and blood samples for translational research;
17. Before patient registration/randomization, written informed consent must be given according to International Conference on Harmonization (ICH)/ Good Clinical Practice (GCP), and national/local regulations.

Exclusion Criteria:

1. Floor-of-mouth primaries or extension onto the floor-of-mouth;
2. Documented evidence of distant metastases (M1) based on a diagnostic, contrast-enhanced whole-body PET-CT scan ;
3. Any previous anti-cancer therapy for HNSCC (surgery, chemo, radiotherapy or molecularly targeted therapy);
4. History of another primary malignancy with the exception of:

   * Malignancy treated with curative intent and with no known active disease ≥2 years before enrolment and of low potential risk for recurrence
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
   * Adequately treated carcinoma in situ without evidence of disease;
5. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study;
6. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before enrolment in the trial;
7. Known contraindication to imaging tracer or nay product of contrast media, or MRI contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) | Day 30 (+5)
  Assessment of the effect of neoadjuvant DaRT on Major Pathological Response following DaRT seeds insertion

SECONDARY OUTCOMES:
Pathological Response | Day 30 (+5)
  Assessment of the effect of neoadjuvant DaRT on pathological response, using a four-point scale following DaRT seeds insertion
Radiological Response | Day 30 (+5)
  Assessment of the effect of neoadjuvant DaRT on radiological response, as measured by the overall response rate (ORR) of the primary tumor and nodes by RECIST 1.1 (based on CT). Each patient will be assigned one of the following categories based on local assessment: complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), early death or not evaluable.
Metabolic Response | Day 30 (+5)
  Assessment of the effect of neoadjuvant DaRT on radiological response, as measured by Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST - based on positron emission tomography (PET-CT)). Each patient will be assigned one of the following categories based on local assessment: complete metabolic response, partial metabolic response, stable metabolic disease, progressive metabolic disease, early death or not evaluable.
Overall Survival (OS) | Up to 24 months
  Defined as the time interval between the date of of DaRT seeds insertion and the date of death for any cause.
Disease Free Survival (DFS) | Up to 24 months
  Defined as time from DaRT seeds insertion to date of first occurrence of any loco-regional progression or recurrence, metastatic progression, or death due to any cause, whichever comes first.
DaRT Safety | From enrolment until 90 days after completion of post-operative treatment
  Measured by the incidence of all adverse events assessed according to CTCAE version 5
Positive Margin Rate | Day 30 (+5)
  Each patient undergoing surgery will be assigned one of the following categories based on the margin in the primary specimen (final margin after resection, if any): positive margin, close margin, clear margin.
Post-operative complications Classification | Day 30 (+5)
  The Clavien-Dindo Classification of Surgical Complications (2009) will be used to grade the complications from I (any deviation from the normal post-operative course without the need for pharmaceutical treatment or surgical, endoscopic, and radiological interventions) to V (Death).

CONTACTS AND LOCATIONS:
Overall Officials: Aron Popovtzer, MD, Principal Investigator — Sharett institute, Hadassah Medical Center - Ein-Kerem
Locations (1):
- Sharett institute, Hadassah University Hospital - Ein-Kerem, Jerusalem, Israel